CLINICAL TRIAL: NCT01240707
Title: Pathophysiologic Changes in the Respiratory System After Fire Smoke Inhalation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Espen Rostrup Nakstad, MD, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: REK S-O, Ref 2010/1340, part A
Record Dates: First submitted 2010-11-10; First posted 2010-11-15 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Bronchial Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LF tests, Fiberoptic bronchoscopy (Other): Spirometry, Peak Expiratory Flow (PEF). Bronchoscopic assessment of soot in central airways.
  Interventions: Other: Fiberoptic bronchoscopy

INTERVENTIONS:
Other: Fiberoptic bronchoscopy — Fiberoptic bronchoscopy performed to remove secretions and assess soot in central airways
  Other Names: Bronchopscopy

SUMMARY:
Fire smoke inhalation may contribute to intrabronchial inflammation, airway obstruction and impaired gas exchange. In this study the investigators will examine if the scope of inhalation injury can be assessed soon after hospital admission based on clinical markers, biochemical markers, Peak Expiratory Flow (PEF), spirometry and bronchoscopy. At 6 months a lung function test and metacholine test will be performed to examine whether patients have developed increased bronchial hyperreactivity (asthma) or not after the initial fire smoke exposure.

DETAILED DESCRIPTION:
Fire smoke inhalation may contribute to intrabronchial inflammation, airway obstruction and impaired gas exchange. The scope of injury in fire smoke victims ranges from cough and minor airway irritation to severe respiratory failure and long term mechanical ventilation in the Intensive Care Unit. Some patients with high HbCO-levels are also treated with hyperbaric oxygen therapy.

In this study the investigators will examine if the scope of inhalation injury can be assessed soon after admission based on clinical markers, biochemical markers, Peak Expiratory Flow (PEF), spirometry and bronchoscopy. The clinical effect of fiberoptic bronchoscopy after severe smoke inhalation will also be examined. At 6 months a lung function test and metacholine test will be performed to examine whether they have developed asthma/increased bronchial hyperreactivity or not after the initial fire smoke exposure. Lab staff (flowcytometer and cytokine analysis) are unaware of patient identity and whether the patient is a smoke-exposed patient or a healthy volunteer in the control group of non-exposed persons.

ELIGIBILITY:
Inclusion Criteria:

* fire smoke exposed patient
* > 18 years of age
* admitted to hospital

Exclusion Criteria:

* < 18 years of ager
* trauma patient

Control group (healthy volunteers/hospital staff):

* > 18 years of age
* non-smoker
* no exposure to fire smoke

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-11; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Positive metacholine test (bronchial hyperreactivity). | 6 months
  At 6 months a lung function test and metacholine test will be performed to examine whether patients have developed asthma/increased bronchial hyperreactivity after the initial fire smoke exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Espen R Nakstad, MD, Principal Investigator — Oslo University Hospital - Ulleval, Norway; Helge Opdahl, MD, PhD, Study Director — Ullevaal University Hospital
Locations (1):
- Oslo University Hospital - Ulleval, Oslo, Oslo County, Norway

IPD SHARING:
Plan to Share IPD: Undecided